CLINICAL TRIAL: NCT02286102
Title: A Prospective Randomized Study on the Clinical Benefits of OrthoPAT Drains for Adults Undergoing Multilevel Spine Surgery for Deformity
Brief Title: A Prospective Randomized Study on the Clinical Benefits of OrthoPAT Drains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-363
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Spine Deformity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OrthoPAT (Experimental): Patients in the experimental group will receive OrthoPAT drains, which will be used to collect and retransfuse postoperative blood loss. Drains will be removed after 48 hours.
  Interventions: Device: OrthoPAT
- Constavac (Active Comparator): Patients identified as active comparator will receive standard Constavac drains, which will be removed after 48 hours.
  Interventions: Device: Constavac

INTERVENTIONS:
Device: OrthoPAT — OrthoPAT drain to collect and retransfuse postoperative blood loss. Drains will be removed 48 hours postoperatively
  Arms: OrthoPAT
Device: Constavac — Constavac drain to collect postoperative blood loss. Drains will be removed 48 hours postoperatively
  Arms: Constavac

SUMMARY:
The examination of the ability of the OrthoPAT® blood collection device to decrease the transfusion rate and volume of adults undergoing posterior spine surgery for deformity correction of 6 levels or more.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the use of postoperative drains with blood salvage capabilities to determine if they decrease both the volume and rate of allogenic blood transfusion in adult patients undergoing multilevel spine surgery for deformity. In addition, the ability of these drains to decrease the complications that are associated with allogenic blood exposure (postoperative infection, volume overload and transfusion reactions) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

The patient is at least 18 years of age The patient is to undergo posterior spine surgery in the thoracic or lumbar region for deformity correction of greater than 6 levels The patient has signed a patient Informed Consent

Exclusion Criteria:

The patient is less than 18 years of age The patient has a hematologic disorder of any etiology The patient has received active anticoagulant therapy, including aspirin, Plavix, Heparin, Lovenox or Coumadin within one week of admission The patient has a known active infection or malignancy. The patient has a terminal illness with a life expectancy of less than one year.

The patient requires immuno-suppressive therapy. The patient is undergoing a combined anterior/posterior fusion. The patient has a history of drug or alcohol abuse that may interfere with his/her ability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Ross, RN, Study Director — Hospital for Special Surgery, New York; Han Jo Kim, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- The Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Constavac | OrthoPAT
Started | 36 | 34
Completed | 35 | 33
Not Completed | 1 | 1
Not completed — Screen Failure | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Constavac | OrthoPAT | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 33 | 68
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 28 | 54
  Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Volume of Allogenic Blood Transfused Postoperatively
Description: The total volume of allogenic blood transfused postoperatively will be measured during the first 48 hours postoperatively while the drains are in place.
Time Frame: 48 hours postoperative
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Constavac | OrthoPAT
Number analyzed (Participants) | 35 | 33
mL | 458.33 (4.28) | 382.35 (62.22)

2. Secondary Outcome: Hemoglobin Levels, Post-Op Day 3
Description: Hemoglobin levels will be measured post-operatively day 3
Time Frame: 3 days postop
Measure: Mean (Standard Deviation); unit: g/Dl (grams/deciliter)
Arm/Group | Constavac | OrthoPAT
Number analyzed (Participants) | 35 | 33
g/Dl (grams/deciliter) | 9.07 (.79) | 9.9 (.99)

3. Secondary Outcome: Hemoglobin Levels, Post-Op Day 2
Description: Hemoglobin levels will be measured post-operatively day 2
Time Frame: 2 days postop
Measure: Mean (Standard Deviation); unit: g/Dl (grams/deciliter)
Arm/Group | Constavac | OrthoPAT
Number analyzed (Participants) | 35 | 33
g/Dl (grams/deciliter) | 9.33 (.88) | 10.19 (1.24)

ADVERSE EVENTS:
Time Frame: From time of surgery to post-op day 3.
Arm/Group | OrthoPAT | Constavac
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes